CLINICAL TRIAL: NCT02300454
Title: Effect of Combination of Non-sLip Element Balloon (NSE) and druG-coated bAlloon (DCB) for In-steNT Restenosis Lesions
Acronym: ELEGANT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mitsui Memorial Hospital (Other)
Collaborators: Teikyo University (Other); Tokai University (Other)
Responsible Party: Principal Investigator, Jiro Aoki, Associate Director, Division of Cardiology, Mitsui Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC2014-14
Record Dates: First submitted 2014-11-14; First posted 2014-11-25 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Coronary Restenosis
Keywords: in-stent restenosis; percutaneous coronary intervention; balloon
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-slip element balloon (NSE) (Active Comparator): Lacrosse® NSE dilatation before use of SeQuent® Please drug coated balloon (DCB)
  Interventions: Device: Non-slip element balloon (NSE)
- Balloon (Placebo Comparator): Non-compliant balloon dilatation before use of SeQuent® Please drug coated balloon (DCB)
  Interventions: Device: Balloon

INTERVENTIONS:
Device: Non-slip element balloon (NSE) — Lacrosse® NSE and SeQuent® Please drug coated balloon (DCB)
  Arms: Non-slip element balloon (NSE)
Device: Balloon — Non-compliant balloon and SeQuent® Please drug coated balloon (DCB)
  Arms: Balloon

SUMMARY:
Use of SeQuent® Please drug coated balloon (DCB) is effective to treat patients with in-stent restenosis (ISR). However, whether the type of pre-dilatation balloon prior to DCB dilatation impacts on clinical and angiographic outcomes or not is unknown. Lacrosse® Non-slip element balloon (NSE) is a balloon catheter with 3 longitudinal plastic elements which are attached to proximal and distal balloon edges. NSE is developed to incise neointimal tissue and avoid balloon slippage without vitiating balloon derivability and crossability. We investigated angiographic and clinical outcomes following normal non-compliant balloon or NSE dilatation prior to DCB dilatation in ISR lesions.This study is a single blinded, multicenter, randomized trial. Total 200 patients with ISR are randomly assigned to treat with non-compliant balloon or NSE before DCB dilatation. Optical coherence tomographic (OCT) analysis are performed before pre-dilatation and after DCB dilatation Follow-up angiography analysis are planned at 8 months in all patients. Clinical follow-up is planned at 8 and 24 months.Primary endpoint is angiographic in-segment late loss at 8 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with in-stent restenosis lesions who are planned to be treated with drug coating balloon

Exclusion Criteria:

* ST elevation myocardial infarction
* stent thrombosis
* severe renal dysfunction (eGFR <30 ml/min) except dialysis
* pregnancy
* planned surgery within 3 months
* shock vital

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2015-06; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Angiographic in-segment late loss | 8 months

SECONDARY OUTCOMES:
angiographic minimal lumen diameter | 8 months
minimal lumen area (OCT analysis) | within one day
mean neointimal area (OCT analysis) | within one day
angiographic acute gain | within one day
Target vessel failure | 8 months and 24 months
  cardiac death, myocardial infarction, target vessel revascularization
the prevalence of stent implantation | within one day
the prevalence of balloon slipping | within one day
  more than 3 mm balloon slipping
DCB length | within one day

OTHER OUTCOMES:
angiographic in-segment late loss | 8 months
  subanalysis: drug eluting stent restenosis
angiographic in-segment late loss | 8 months
  subanalysis: slipping group
angiographic in-segment late loss | 8 months
  subanalysis: diffuse, occlusive, and proliferative restenosis type
angiographic in-segment late loss | 8 months
  subanalysis: in-stent re-restenosis lesion
angiographic in-segment late loss | 8 months
  subanalysis: stent diameter 2.25 or 2.5 mm

CONTACTS AND LOCATIONS:
Overall Officials: Ai Teramoto, Study Director — Teikyo Academic Research Center
Locations (2):
- Japan (2):
  - Tokai University, Isehara, Kanagawa
  - Mitsui Memorial Hospital, Chiyoda-Ku, Tokyo

REFERENCES:
- [Derived] Aoki J, Nakazawa G, Ando K, Nakamura S, Tobaru T, Sakurada M, Okada H, Hibi K, Zen K, Ikuta A, Fujii K, Habara M, Ako J, Asano T, Ozaki S, Fusazaki T, Kozuma K; ELEGANT investigators. Impact of hemodialysis on clinical and angiographic outcomes in in-stent restenotic lesions following optical coherence tomography-guided drug-coated balloon treatment. Cardiovasc Interv Ther. 2021 Oct;36(4):429-435. doi: 10.1007/s12928-020-00718-7. Epub 2020 Oct 13. PMID 33048289